CLINICAL TRIAL: NCT04139915
Title: A Multicenter, Randomized, Double Blind, Placebo-Controlled, Phase 3 Study to Determine if RTB101 Prevents Clinically Symptomatic Respiratory Illness in the Elderly
Brief Title: Effect of RTB101 on Illness Associated With Respiratory Tract Infections in the Elderly
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Phase 3 trial RTB-101-204 study did not meet its primary endpoint
Sponsor: Restorbio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RTB-101-205
Record Dates: First submitted 2019-10-17; First posted 2019-10-25 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Clinically Symptomatic Respiratory Illness
Keywords: Mechanistic Target of Rapamycin (mTOR); Influenza; Virus; Pneumonia; Immunosenescence; Respiratory Tract Infections
MeSH Terms: conditions — Hereditary Sensory and Autonomic Neuropathies; Influenza, Human; Virus Diseases; Pneumonia; Respiratory Tract Infections | interventions — dactolisib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 10 mg daily RTB101 (Experimental): Oral RTB101 10 mg hard gelatin capsule once daily for 16 weeks
  Interventions: Drug: Dactolisib
- Placebo (Placebo Comparator): Oral matching placebo once daily for 16 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dactolisib — TORC1 inhibitor
  Other Names: RTB101; BEZ235
  Arms: 10 mg daily RTB101
Drug: Placebo — Placebo capsule
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if RTB101 prevents illness associated with respiratory tract infections in people ≥65 years of age.

DETAILED DESCRIPTION:
RTB-101-205 is a randomized, double-blind, placebo-controlled, multicenter, parallel-group, Phase 3 study to determine if RTB101, a selective TORC1 inhibitor, prevents illness associated with respiratory tract infections (defined as clinically symptomatic respiratory illness) in adults ≥65 years of age. This trial is being conducted in follow up to two Phase 2 trials in older adults in which RTB101 10 mg administered once daily for up to 16 weeks during winter cold and flu season was observed to reduce the incidence of respiratory illness associated with respiratory tract infections.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be ≥65 years of age
* Subjects should require no or minimal assistance with self-care and activities of daily living. Subjects in assisted-living or long-term care residential facilities that provide minimal assistance are eligible
* Sexually active male subjects with a partner of child-bearing potential must be willing to wear a condom while on study drug and for 1 week after stopping study drug and should not father a child in this period

Exclusion Criteria:

* Subjects who are current smokers, stopped smoking ≤ 1 year prior to screening, or have and a ≥ 10 pack year smoking history
* Subjects with a medical history of clinically significant lung diseases (including COPD) other than asthma
* Subjects with current evidence of a serious and/or unstable medical disorder
* Subjects with unstable cardiac conditions
* Subjects with a history of systemic autoimmune diseases
* Subjects with Type I diabetes mellitus
* Subjects with a history of immunodeficiency diseases, including a positive human immunodeficiency virus (HIV) test result
* Infection with Hepatitis B (HBV) or Hepatitis C (HCV)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10-21 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with clinically symptomatic respiratory illness | Through Week 16

SECONDARY OUTCOMES:
Percentage of subjects with clinically symptomatic respiratory illness associated with ≥1 laboratory-confirmed pathogen(s) | Through Week 16
Rate of clinically symptomatic respiratory illness (with or without an associated laboratory-confirmed pathogen) | Through Week 16
Rate of clinically symptomatic respiratory illnesses associated with ≥1 laboratory-confirmed pathogen(s) | Through Week 16
Time to alleviation of moderate and severe respiratory illness symptoms due to clinically symptomatic respiratory illness | Through Week 16
Percentage of subjects with severe respiratory illness symptoms due to clinically symptomatic respiratory illnesses | Through Week 16
Number of participants with treatment-emergent adverse events as assessed by CTCAE v5.0 | Through Week 20
Rate of clinically symptomatic respiratory illnesses associated with specific laboratory-confirmed viruses | Through Week 16
  Descriptive statistics will be provided for the rate of clinically symptomatic respiratory illnesses associated with specific laboratory-confirmed viruses. No formal statistical tests will be conducted.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Restorbio Inc.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mannick JB, Morris M, Hockey HP, Roma G, Beibel M, Kulmatycki K, Watkins M, Shavlakadze T, Zhou W, Quinn D, Glass DJ, Klickstein LB. TORC1 inhibition enhances immune function and reduces infections in the elderly. Sci Transl Med. 2018 Jul 11;10(449):eaaq1564. doi: 10.1126/scitranslmed.aaq1564. PMID 29997249